CLINICAL TRIAL: NCT06077799
Title: prehospItal maNagement oF paroxysmaL supraventrICular Tachycardia - Gestione Preospedaliera Della Tachicardia Parossistica Sopraventricolare
Brief Title: prehospItal maNagement oF paroxysmaL supraventrICular Tachycardia
Acronym: INFLICT
Status: Completed | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Azienda Regionale Emergenza Urgenza - AREU Lombardia (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Sponsor
Other Study IDs: 296-2023-OSS-AUSLBO
Record Dates: First submitted 2023-07-10; First posted 2023-10-11 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Tachycardia, Supraventricular
Keywords: supraventricular tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- supraventricular tachycardia treated with intra-venous adenosine: supraventricular tachycardia treated with intra-venous adenosine
- supraventricular tachycardia treated with electrical synchronised cardioversion: supraventricular tachycardia treated with electrical synchronised cardioversion

SUMMARY:
Retrospective multicentre study on management of supraventricular tachycardia in prehospital setting.

DETAILED DESCRIPTION:
Supraventricular tachycardia in prehospital setting may be managed with adenosine administration or with synchronised electrical cardioversion and there's no clear advantage between the two, even if international guidelines suggests to practice drug-first method.This study aims to evaluate any difference in outcomes and efficacy of the two methods and possible adverse effects of both.

ELIGIBILITY:
Inclusion Criteria:

* patients accepting to participate
* patients affected by supraventricular tachycardia that are managed prehospitally by the emergency medical service

Exclusion Criteria:

* not willing to participate, not able to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients affected by any form of supraventricular tachycardia
Sampling Method: Non-Probability Sample
Enrollment: 1234 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of adenosine versus electric cardioversion in obtaining successful cardioversion of PSVT | Prehospital EMS assistance time
  absolute numbers and relative percentages of successful prehospital cardioversions obtained with the two techniques

SECONDARY OUTCOMES:
diagnostic accuracy for supraventricular tachycardia of the emergency medical service personnel | Prehospital EMS assistance time
  Sensitivity for PSVT of the EMS personnel
adverse events | Prehospital EMS assistance time
  incidence of predefined serious adverse events (SAE) between the two groups

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Unità Sanitaria Locale, Bologna, Bologna
  - Agenzia Regionale Emergenza Urgenza (AREU), Dipartimento di Emergenza e Accettazione, ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy
  - Azienda Ospedaliera Universitaria Maggiore della Carità, Novara, Italy, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gamberini L, Carinci V, Pallavicini P, Rovera M, Tartaglione M, Gioachin R, D'ambrosio A, Fiameni R, Baroncini S, Allegri D, Coniglio C, Semeraro F, Ristagno G; INFLICT working group. Prehospital management of supraventricular tachycardia: a multicentre study of current practices with a subgroup propensity score-based comparison of adenosine and electrical cardioversion in unstable patients. Resuscitation. 2025 Oct;215:110707. doi: 10.1016/j.resuscitation.2025.110707. Epub 2025 Jul 7. PMID 40633750